CLINICAL TRIAL: NCT06969560
Title: There's No Place Like Home…Feasibility of Remote Physiological Monitoring in Childhood Heart Failure
Brief Title: WeRoaM: Wearable Remote Monitoring in Heart Failure
Acronym: WeRoaM:
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Pro00126084
Record Dates: First submitted 2025-04-22; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: remote physiologic monitoring; heart failure; at-risk; telemonitoring technology; pediatric
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- paediatric outpatients (8 to 18 years old) with diagnosis of cardiomyopathy: This study will enroll 100 paediatric outpatients (8 to 18 years old) with diagnosis of cardiomyopathy (with systolic or diastolic dysfunction), subjects with congenital heart disease with biventricular or univentricular physiology plus systemic ventricular dysfunction from 4 tertiary heart failure care centres.
  Patients will participate in a remote physiologic monitoring program using bluetooth enabled devices for 12 weeks. Devices as part of the study intervention include: Skiin chest band and ECG device; blood pressure monitor; pulse oximeter; weight scale.
  Interventions: Device: Remote Physiologic Monitoring (RPM)

INTERVENTIONS:
Device: Remote Physiologic Monitoring (RPM) — The intervention consists of a remote physiologic monitoring (RPM) program which makes use of a wearable Skiin chest band and ECG device, a blood pressure monitor, a pulse oximeter, and a weight scale; the RPM program will occur for 12 weeks Participants will wear the Skiin device continuously for the first 48-hours and then for a 12-hour span each day following that. Participants will measure their blood pressure, oxygen saturation, and weight once a day for the full 12 weeks.

SUMMARY:
Remote physiologic monitoring (RPM) of heart failure (HF) patients with a virtual platform is well established in adult care. However, this technology remains untested in pediatrics and care continues to rely on a hospital-based model which presents challenges in providing equitable access to care for those with lower socio-economic status or living remotely. Telemonitoring technology tailored for children with machine-based algorithms to predict deterioration is needed to facilitate the equitable provision of safe, home-based care, especially in vulnerable populations.

This study will enroll 100 pediatric outpatients with or at risk of deteriorating HF from 4 tertiary pediatric heart failure care centres in Canada. We will use a wearable Bluetooth enabled textile (Skiin device), developed by Myant Inc (Toronto, ON), that can monitor heart rate, heart rhythm, respiratory rate and activity, together with additional home-based monitoring of blood pressure (BP), oxygen saturations and weight. The smart textile will be paired to an RPM platform, SphygmoTM (mmHG Inc).

The goal of this project is to assess the feasibility and acceptability of RPM in pediatrics and validate a RPM-based risk prediction model for pediatric HF patients.

DETAILED DESCRIPTION:
Remote physiologic monitoring (RPM) refers to utilizing non-invasive medical devices to obtain physiologic data, such as pulse oximetry, blood pressure, weight, and electrocardiography at home. Recent advances in RPM have facilitated improved home-based care, reduced hospitalizations, and improved quality of life in adult heart failure populations. Additionally, the integration of multiple physiologic variables acquired through remote physiologic monitoring into machine learning algorithms has been shown to predict hospitalization for heart failure. Previous paediatric studies have demonstrated the utility of incorporating multiple physiologic variables into risk prediction algorithms for cardiac events. This is particularly important in heart failure cohorts where limits of acceptability are often nuanced and patient specific. The use of multiple physiologic parameters creates a more comprehensive insight into the complex pathophysiologic changes in heart failure.

However, the use of RPM devices in children remains limited due to a lack of validated devices and uncertainty about the acceptability and uptake of such interventions. This is partly due to challenges developing devices that can be easily applied, and digital platforms suited to the wider range and variability in body sizes and physiologic parameters. Thus, care of children with heart failure continues to rely on hospital-based models, where tertiary heart failure centers serve large geographically and socio-economically diverse populations. A validated paediatric virtual home monitoring system using RPM to predict clinical deterioration could safely facilitate earlier discharge, reduce the need for outpatient hospital visits, and potentially improve outcomes while minimizing family social disruption and school absence.

The overarching goal of this project is to assess the feasibility of RPM in paediatrics and validate a RPM based risk prediction model for paediatric patients with or at-risk of heart failure, with a view to facilitating safe home-based care across geographically and socially diverse urban, rural, and remote communities. To achieve this goal, this study proposes to utilize a wearable Bluetooth enabled textile (Skiin Device) that can monitor heart rate and rhythm, respiratory rate and activity, together with additional home-based monitoring of blood pressure, oxygen saturations and weight. The textile, developed by Myant (Toronto, ON) has completed pilot testing at SickKids to assess its validity in an outpatient setting (NCT04305340). The Skiin textile will be paired to its software solution, the Myant Health Platform (MHP), which comprises the Skiin Connected Life App (phone application), the Myant Back End (cloud storage of data) and the Myant Virtual Clinical Portal (internet browser visualization of data collected). The Skiin Connected Life App will be used for collection of ECG, heart rate, body temperature, and physical activity throughout the day, and can generate the following average metric for each night when the device is used: resting heart rate, respiratory rate, resting heart rate variability, sleep duration, body temperature.

The MHP will be paired with another RPM platform, SphygmoTM (mmHG Inc). The Sphygmo™ platform consists of a smartphone App (Android, iOS), which can be linked with Bluetooth-compatible devices for automated uploading of measurements to a clinician portal. This platform, originally developed for adults, has the ability to connect with blood pressure, heart rate, weight, and oxygen saturation devices. This platform will be used for collection of additional physiologic data as above and is currently under study at Stollery Children's Hospital. The two systems will have a single-sign on feature allowing their integrated use by the patient, their families, and the research team. We will leverage descriptive and predictive analytics to augment clinician monitoring by defining trajectories and longitudinally predicting risk of key adverse outcomes.

Study Objectives Primary Objectives

1. To investigate the feasibility of a remote physiological monitor using a textile smart garment (Skiin devices) using the Skiin Connected Life App along with additional standard home monitoring tools (BP monitor, weigh scales) that are paired with a Bluetooth enabled app (SphygmoTM)
2. To test the acceptability of a remote physiological monitor using a textile smart garment (Skiin devices) along with the acceptability of a Bluetooth enabled app (SphygmoTM)

Secondary Objectives

1. To leverage analytical methods to develop descriptive and predictive tools using RPM that augment detection of clinical deterioration in pediatric patients as measured by admission, adverse cardiac events and patient reported outcomes within 6-months post intervention.

Study Duration: Patients will be recruited over a 2-year period.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 8-18 years of age who are outpatients at time of study enrollment.
* Patients with a chest size of at least 69.85 cm in perimeter/circumference (as measured under the pectoral muscles)
* Patients at-risk for heart failure and with American Heart Association (AHA) Stage B-D Heart Failure will be included in this study irrespective of heart failure medication use.
* HF etiologies include: congenital cardiac malformation with systemic ventricular systolic dysfunction, idiopathic cardiomyopathy, familial/inherited and/or genetic cardiomyopathy, history of myocarditis with persistent ventricular dysfunction, neuromuscular disorder, inborn error of metabolism, mitochondrial disorder, acquired (chemotherapy, iatrogenic, infection, rheumatic, or nutritional), ischemic (e.g., Kawasaki disease and post-operative HF), and left ventricular non-compaction, restrictive cardiomyopathy and HCM with systolic or diastolic dysfunction.

Exclusion Criteria:

* Patients within 3 months of a surgery.
* Patients supported by ventricular assist device at study onset.
* Inability to use technology due to physical or cognitive impairment in the patient or caregiver.
* Non-English speaking.
* Patients who have an implantable cardiac defibrillator or pacemaker
* Patients whose chest size is too large or small to fit available sizes of the Skiin device.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will enroll 100 paediatric outpatients (8 to 18 years old) with diagnosis of cardiomyopathy (with systolic or diastolic dysfunction), subjects with congenital heart disease with biventricular or univentricular physiology plus systemic ventricular dysfunction from 4 tertiary heart failure care centres.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Remote Physiologic Monitoring (RPM) Program- Recruitment | 2 years
  Feasibility will be assessed by recruitment rates (the number of participants recruited
Feasibility of Remote Physiologic Monitoring (RPM) Program- Retention | 2 years
  Feasibility will be assessed by retention rate (the number of participants who complete measures at baseline and at follow up post intervention)
Feasibility of Remote Physiologic Monitoring (RPM) Program- Access | 2 years
  Feasibility will be assessed by the percentage of people with access to Wi-Fi and smart device
Acceptability of Remote Physiologic Monitoring (RPM) Program | 2 years
  Acceptability will be assessed by compliance defined as >80% of the physiologic monitoring requested has been captured twice daily for a period of 12 weeks; completion of the Medtech 20 questionnaire will also inform on acceptability.

SECONDARY OUTCOMES:
Composite End-Point Assessing Remote Physiologic Monitoring (RPM) Program | 2 years
  For the secondary outcome we will use a composite end-point. Given the low prevalence and rarity of events such as death or transplant from chronic heart failure in paediatrics, there is limited potential for large outcome trials. As a result, we will use a composite end-point designed for the PANORAMA-HF study and based on Packer's composite score which has been extensively used in adult heart failure studies.
  Patients will be ranked within 5 categories from worst to best based on heart failure events such as death, transplant listing, need for mechanical circulatory supports, as well as progression of heart failure symptoms by NYHA or Ross Class and patient reported outcomes as assessed by the PedsQL and PGIS. Patients who experience a clinical event during follow up will be classified into category 1 and 2. Patients without a clinical event during follow up will be divided into 3, 4 and 5 based on change from baseline symptoms and functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Conway, MD, MSc, Principal Investigator — University of Alberta/Stollery Children's Hospital; Aamir Jeewa, MD, Principal Investigator — University of Toronto; The Hospital for Sick Children
Locations (4):
- Canada (4):
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy and confidentiality, no IPD will be shared. Only group trends will be reported.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT06969560/Prot_SAP_000.pdf